CLINICAL TRIAL: NCT03044990
Title: Study on the Prognosis of Patients With Acute Coronary Syndrome Complicated With Renal Insufficiency: a Prospective, Multicenter, Observational Study
Brief Title: Prognosis of Patients With Acute Coronary Syndrome Complicated With Renal Insufficiency(PACS-RI)
Acronym: PACS-RI
Status: Completed | Type: Observational
Sponsor: Henan Institute of Cardiovascular Epidemiology (Other)
Responsible Party: Sponsor
Other Study IDs: HenanICE201603
Record Dates: First submitted 2017-01-19; First posted 2017-02-07 (Estimated); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Acute Coronary Syndrome
Keywords: Acute coronary syndrome; renal insufficiency; mortality
MeSH Terms: conditions — Acute Coronary Syndrome; Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Several epidemiologic studies reported that patients with renal insufficiency might have increased cardiovascular disease-related mortality rates after Percutaneous coronary intervention (PCI) . The increased risk in this population may be related to the less use of standard guideline-based treatment and the resulting inability to perform PCI effectively. Recently, with the technology improvement and the progress in clinical trials, Chinese guidelines have made new recommendations about the patients with acute coronary syndrome(ACS) in different states of renal function. However, scant epidemiologic information exists on the prognosis of those patients, especially in Henan. And there is still some uncertainty whether those patients are using the latest guideline recommended treatment.

This multicenter, prospective, observational study is aimed to evaluate the long prognosis in patients with acute coronary syndrome complicated with renal insufficiency, and to analysis its related factors that influence the outcomes.

DETAILED DESCRIPTION:
1. Henan institute of cardiology epidemiology is responsible for design, data quality control and statistical analysis.
2. Data were collected using a uniformed Case Report Form(CRF) by trained staff at each hospital.
3. Sample size estimation: Based on retrospective observational cohort of ACS patients, 1-year mortality in normal renal function and renal disfunction were 2.8% and 7.9%, respectively. To achieve a precision of 15% with an α of 0.05, the loss ratio of following-up is 10%.The investigators would need a sample of 2000.
4. Statistical analysis plan: the investigators will report summary statistics for patient characteristics, renal function status, comorbidities, treatment strategies and outcomes. the investigators will also undertake the following prespecified subgroup analyses: age, sex, STE-ACS or NSTE-ACS, history of diabetes, history of hypertension, smoking and Syntax score.
5. Quality assurance plan 1)Diagnosis of ACS is according to the third universal definition.2)Before registry, a training program on study objectives, data collection, and ACS management is given to the primary investigator and related staff at each participating center.3)Henan institute of cardiology epidemiology will regularly monitored at least 10% of CRFs for accuracy against medical records. If the CRFs are not completed with 98% accuracy, all CRFs are considered unqualified and this staff will be retrained.4)Before entering into the computer, data is queried for invalid and illogical values by research staff in Henan institute of cardiology epidemiology. Participating centres who has the high error rate of data, and no change in 6 months shall be deemed abandoned automatically; participating centres who has the high quality of data will be issued a certificate to reward.5)Investigator meeting will be annually held to conclude the progress, solve existing problems and strengthen program training.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years.
2. Patients with clinical evidence of acute coronary syndrome, including ST segment elevation myocardial infarction (STEMI), non ST segment elevation myocardial infarction (NSTEMI) and unstable angina.
3. Informed consent signed by patients or legal guardians.

Exclusion Criteria:

1. Non-atherosclerotic coronary heart disease
2. Organ failure other than heart failure and kidney failure
3. Considered not fit for the study due to other reasons, including but not restricted to : a. Severe infection; b. cachexia;c.maintenance hemodialysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 7 eligible sites in Henan province will participate. Each site will enroll patients who meet the inclusion criteria consecutively.
Sampling Method: Probability Sample
Enrollment: 2014 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiovascular and cerebrovascular events | 1 year
  including all-caused death, nonfatal- myocardial infarction,and stroke

SECONDARY OUTCOMES:
Major adverse cardiovascular and cerebrovascular events | At discharge(an average of 10 days),6 month
  including all-caused death, nonfatal- myocardial infarction,and stroke
Coronary revascularization | 6 month,1 year
Re-hospitalized | 6 month,1 year
Renal-Replaced therapy | At discharge(an average of 10 days),6 month,1 year
Bleeding according to GUSTO bleeding grade(excluding hemorrhage stroke) | At discharge(an average of 10 days),6 month,1 year
Cardiogenic shock | At discharge(an average of 10 days)
New arrhythmia | At discharge(an average of 10 days)

CONTACTS AND LOCATIONS:
Overall Officials: Chuanyu Gao, MD, Principal Investigator — Henan Institute of Cardiovascular Epidemiology
Locations (1):
- Henan province people's hospital, Zhengzhou, Henan, China